CLINICAL TRIAL: NCT06535477
Title: Fall Risk Assessment With an Innovative Device for Quantifying Gait and Static Balance in Geriatric Consultation
Acronym: PARACHUTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A00055-42
Record Dates: First submitted 2024-06-24; First posted 2024-08-02 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Risk of Falling in the Elderly
Keywords: Falls; static balance; Spatio temporal parameters

STUDY DESIGN:
Intervention Model Description: Assessing frailty in elderly patients using Fried Frailty and "Short Emergency Geriatric Assessment" scales combined with measurement - via the AbilyCare device - of the two markers of balance and gait
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Fall risk assessment — Assessing frailty in elderly patients using Fried Frailty and "Short Emergency Geriatric Assessment" scales combined with measurement - via the AbilyCare device - of the two markers of balance and gait

SUMMARY:
The main objective of this monocentric, non-randomized, prospective study was to evaluate the predictive capacity of a balance score based on spatio-temporal parameters of postural balance.

DETAILED DESCRIPTION:
Patient recruitment will take place at one center. The inclusion period is 6 months and the participation period for each subject will be 12 months with 3 visits: initial visit, telephone visit at 6 months, M12 consultation visit, and the end-of-study visit.

Consent will be obtained prior to participation, and the following data will be collected during the visits: Demographic data (age, gender), weight, height, geriatric assessment. Current treatment (molecules, date of introduction, dosage). Biological data: Albumin, Pre-Albumin, Creatinine, Hemoglobin, Vitamin D.

Static balance parameters via AbilyCare (static balance test, inspired by the Romberg test, on a balance platform, 30 seconds eyes open then 30 seconds eyes closed).

The total duration of the research is 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject with a "Autonomie, Gérontologie, Groupes IsoRessources" (GIR) score ≥ 4 at the time of consultation
* Subject presenting an The mini mental status exam (MMSE) score ≥ 18 at the time of consultation
* Subject agreeing in writing (consent), after having been informed and given a reasonable period of reflection, to participate in the study
* Subject affiliated to a social security scheme.

Exclusion Criteria:

* Subjects with a major or systemic pathology likely to significantly impair motor skills (inability to perform a 10m walking test without assistance, inability to perform a balance test on a scale without assistance (30 seconds eyes open / 30 seconds eyes closed),
* Subject with an advanced neurodegenerative pathology (Alzheimer, Parkinson, etc.) deemed incompatible with the objectives of the study by the investigator,
* Subjects with a history of disabling cerebrovascular accident,
* Subject with an active disabling cancer,
* Subjects with severe psychiatric disorders affecting their ability to perform walking and balance tests and/or answer study questionnaires,
* Subjects benefiting from a technical aid for walking and balance such as a cane, walker, etc. (only orthopedic insoles and shoes are accepted); subjects with a total hip or knee prosthesis are included,
* Subject having been hospitalized for a fall in the last 3 months prior to inclusion,
* Subject unable to understand the purpose of the research, answer questions and give his/her decision to participate in the study,
* Subject already included in another research study involving the human body,
* Subject not affiliated to a social security scheme or not benefiting from such a scheme.
* Person deprived of liberty by judicial or administrative decision
* Person of full age subject to a legal protection measure (guardianship, curatorship, safeguard of justice) or unable to express consent.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 169 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
Balance score | 12 months
  The balance score, based on a learning model incorporating spatio-temporal parameters of pressure center displacement. These parameters include amplitude along the anterior-posterior and medio-lateral axes, surface area covered, and displacement speed. The overall score is calculated on the basis of model-building data from profiles of people with and without previous falls. This score, evaluated from 0 to 100, indicates the level of balance, with a score of 99 representing optimal balance. The lower the score, the more precarious the balance, thus approximating a potential faller profile.

SECONDARY OUTCOMES:
Evaluation of the association between each static balance indicator and fall occurrence | 12 months
  The following indicators will be analyzed:
  * Oscillation area in mm² : Area covered by the displacement of the center of pressure, calculated by tracing the trajectory of the center of pressure and determining the minimum area that encompasses all these trajectories (contained within an ellipse of 90% confidence).
  * Sway density in seconds : Duration (travel time) during the entire sequence (30s) when the center of pressure remains in the vicinity (radius less than 5 mm) of each calculated point of the center of pressure's position.
  * Lateral variance in mm² : Extent of variability in the position of the center of pressure around an average position on the medial-lateral axis.
  * Average oscillation speed in mm/s : Average speed of displacement of the center of pressure in all directions.

OTHER OUTCOMES:
Measuring cognitive impairment according Mini-Mental State Examination (MMSE) score | 12 months
  The Mini-Mental State Examination is an unabbreviated scale title. This scale was developed as a brief screening tool to provide a quantitative evaluation of cognitive impairment and to record cognitive changes over time.
  The measure yields a total score of 30. A score of 23 or less is the generally accepted cutoff point indicating the presence of cognitive impairment. Levels of impairment have also been classified as none (24-30); mild (18-23) and severe (0-17)
Assessment of physical frailty according Fried scale | 12 months
  This is an unabbreviated scale title.
  Assessment of 5 dimensions:
  * 0, 1 or 2 pathological dimensions = lack of frailty
  * 3, 4 or 5 pathological dimensions = presence of frailty
Assessment of Failty status using the Short Emergency Geriatric Assessment (SEGA) | 12 months
  This is an unabbreviated scale title.
  if SEGA score < ou = 8 : Not very frail if it contained in the interval [9;11] : Rather frail if it > ou = 12 : Very frail
Assessment of the degree of autonomy according AGGIR score | 12 months
  There are six levels of GIR (GIR 1-6):
  * GIR 1-2 correspond to the lowest level of autonomy
  * GIR 3 and 4 correspond to average levels of loss of autonomy
  * GIR 5-6 correspond to the highest level of autonomy

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Pariel, MD, Study Chair — Ambulatory Care Department, Charles Foix Hospital; Lina MICHELET, MD, Study Director — Abilycare
Locations (1):
- Ambulatory Care Department, Charles Foix Hospital, Ivry-sur-Seine, IIe-de-France, France

IPD SHARING:
Plan to Share IPD: No